CLINICAL TRIAL: NCT04514874
Title: Assessment of the Prevalence and the Impact of the COVID-19 Epidemic in the French Flight Crew in 2020
Acronym: Covaé
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-26; 2020-A01459-30 (Other: IDRCB)
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Self-questionnaire about socio-demographical status, health status and lifestyle habits during and following the COVID-19 pandemic.

SUMMARY:
The aeronautical community was also affected and greatly impacted economically and socially by the Covid-19 pandemic. Away from the acute phase, the epidemiological impact and the consequences of this disease within the French aviation flight crew population must be assessed. This study is aimed at providing original epidemiological data among civil and military aircrew, prior to possible prevention strategies or countermeasures to optimize risk management in terms of aviation safety and to promote, if necessary, future targeted studies.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Professional military aircrew
* Presenting himself/herself for a periodic medical exam

Exclusion Criteria:

* Under 18 years of age
* Parachutists
* Non-professional aircrew
* Presenting himself/herself for a first medical exam
* Pregnant woman, parturient, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of professional military aircrew of all aeronautical specialties presenting themselves for a periodic medical exam.
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of COVID-19 infection among French military professional aircrew | At enrollment
  Prevalence of COVID-19 infection will be estimated on the basis of the replies to the questionnaire

SECONDARY OUTCOMES:
Predictive factors of COVID-19 infection | At enrollment
  Predictive factors of COVID-19 infection will be assessed using a top-down logistic regression model taking into account socio-demographic and occupational variables.
Techniques used for COVID-19 screening | At enrollment
  Techniques used for COVID-19 screening will be estimated on the basis of the replies to the questionnaire (among participants who reported being tested for COVID-19)
Reasons for COVID-19 screening | At enrollment
  Reasons for COVID-19 screening will be estimated on the basis of the replies to the questionnaire (among participants who reported being tested for COVID-19)
Experienced symptoms of COVID-19 | At enrollment
  Experienced symptoms of COVID-19 will be estimated on the basis of the replies to the questionnaire (among participants who reported being infected)
Medical care of COVID-19 | At enrollment
  Medical care of COVID-19 will be estimated on the basis of the replies to the questionnaire (among participants who reported being infected)
Social consequences of the COVID-19 pandemic | At enrollment
  Social consequences of the COVID-19 pandemic will be estimated on the basis of the replies to the questionnaire
Factors associated with pejorative consequences of the COVID-19 pandemic | At enrollment
  Factors associated with pejorative consequences of the COVID-19 pandemic will be assessed using a top-down logistic regression model taking into account socio-demographic and occupational variables.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre d'Expertise Medicale du Personnel Navigant (CEMPN) de l'Hôpital d'Instruction des Armées Percy, Clamart
  - Centre d'Expertise Medicale du Personnel Navigant (CEMPN) de l'Hôpital d'Instruction des Armées Sainte-Anne, Toulon

IPD SHARING:
Plan to Share IPD: Undecided